CLINICAL TRIAL: NCT05510245
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL-GROUP STUDY TO EVALUATE THE PHARMACOKINETICS OF PF-07081532 IN ADULT PARTICIPANTS WITH TYPE 2 DIABETES MELLITUS WITH VARYING DEGREES OF RENAL IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT RENAL IMPAIRMENT
Brief Title: A Clinical Trial of the Study Medicine (PF-07081532) in People With Diabetes and Kidney Dysfunction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate clinical development of lotiglipron is based on pharmacokinetic data from Phase 1 drug-drug-interaction studies and laboratory measurements of elevated transaminases in these Phase 1 studies as well as a Phase 2 study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C3991007
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes; Renal Impairment
Keywords: Type 2 Diabetes; Renal impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Participants without renal impairment will receive a single 20 mg dose of PF 07081532, administered orally
  Interventions: Drug: PF-07081532
- Group 2 (Experimental): Participants with mild renal impairment will receive a single 20 mg dose of PF 07081532, administered orally
  Interventions: Drug: PF-07081532
- Group 3 (Experimental): Participants with moderate renal impairment will receive a single 20 mg dose of PF 07081532, administered orally
  Interventions: Drug: PF-07081532
- Group 4 (Experimental): Participants with severe renal impairment will receive a single 20 mg dose of PF 07081532, administered orally
  Interventions: Drug: PF-07081532

INTERVENTIONS:
Drug: PF-07081532 — One PF-07081532 20 mg tablet, administered orally

SUMMARY:
The purpose of this study is to understand the effects of kidney functional impairment may have on the study medicine (PF-07081532). People with certain level of kidney functional impairment may process PF-07081532 differently from healthy people. PF-07081532 is developed as a potential treatment for type II diabetes.

Participants will take the study medicine as a tablet by mouth once at the study clinic and then will stay at the study clinic for about 7 days. During that time, the study team will monitor their treatment experience and take some blood samples to test the level of PF-07081532. This will help us understand if certain degree of kidney functional impairment will have an effect on the study medicine PF-07081532.

ELIGIBILITY:
Inclusion Criteria:

1. Stable renal function (for participants not on dialysis) defined as ≤25% difference between 2 measurements of BSA-unnormalized eGFR
2. A prior diagnosis of T2DM with an HbA1c ≥6% and ≤10.5%
3. Women may be of child-bearing potential
4. BMI of 17.5 to 45.4 kg/m2
5. NORMAL FUNCTION (GROUP 1): Normal renal function (mean eGFR ≥90 mL/min) based on an average of measures from Screening visits S1 and S2 (eGFR should be calculated using the 2021 CKD EPI Scr-Scys combined equation:

   * Demographically comparable to participants with impaired renal function at Screening
   * A body weight within ±15 kg of the mean body weight of the pooled renal impairment groups (Groups 2, 3 and 4)
   * An age within ±10 years of the mean age of the pooled renal impairment groups (Groups 2, 3 and 4)
   * Attempts will be made to ensure that the male to female distribution in Group 1 is comparable to that in the pooled renal impairment groups (Groups 2, 3 and 4).

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus or secondary forms of diabetes, or history of diabetic ketoacidosis.
2. History of myocardial infarction, unstable angina, arterial revascularization, stroke, New York Heart Association Functional Class II-IV heart failure, or transient ischemic attack within 3 months of Screening
3. Personal or family history of MTC or MEN2, or participants with suspected MTC per the investigator's judgement.
4. History of acute pancreatitis within 6 months before Screening or any history of chronic pancreatitis.
5. Urinary incontinence.
6. Participants with acute renal disease.
7. Renal allograft recipients.
8. Participants who have previously received a kidney, liver, or heart transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated due to the termination of clinical development of PF-07081532. As of the last participant last visit (LPLV) date (20 Jul 2023), a total of 18 participants were enrolled at 2 sites in the United States, and no participants without renal impairment were enrolled due to early study termination.
Groups:
- Mild Renal Impairment: Participants with mild renal impairment received a single dose of PF-07081532 20 mg orally.
- Moderate Renal Impairment: Participants with moderate renal impairment received a single dose of PF-07081532 20 mg orally.
- Severe Renal Impairment: Participants with severe renal impairment received a single dose of PF-07081532 20 mg orally.
Period: Overall Study
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 5 | 5 | 8
Completed | 4 | 5 | 8
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 5 | 5 | 8 | 18
Age, Continuous [Median (Full Range); unit: Years] | 68.0 [54 to 83] | 63.0 [55 to 71] | 66.5 [52 to 75] | 66.0 [52 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 2 | 3 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 3 | 1 | 5
  White | 4 | 2 | 7 | 13
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI= {Weight (kilograms [kg])} / {height (centimeters [cm] )*0.01}^2
  kg/m^2 | 29.1 (8.12) | 31.2 (6.89) | 33.7 (7.86) | 31.7 (7.49)
Body Surface Area (BSA)-Unnormalized Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: Milliliters per minute (mL/min)] — BSA-Normalized eGFR was calculated using the 2021 chronic kidney disease epidemiology (CKD-EPI) serum creatinine (Scr) - serum cystatin C (Scys) Combined Equation. Average of the measurements at screening visits S1 and S2 were used in analyses. For participants on dialysis, screening visit S2 was optional. BSA=[weight (kg)^0.425 * height (cm)^0.725]*0.007184. BSA-Unnormalized eGFR=BSA-Normalized eGFR (mL/min/1.73m^2) * [BSA (m^2) /1.73].
  Milliliters per minute (mL/min) | 80.6 (8.26) | 48.7 (6.43) | 15.7 (8.31) | NA (NA) — BSA-unnormalized eGFR is summarized and reported by renal impairment level (ie, mild, moderate, and severe) to show how the values differ across levels of renal impairment. The overall summary for total BSA-unnormalized eGFR is not provided because it is not of interest and not particularly meaningful for overall participants with different levels of renal impairment.

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) for PF-07081532 Following a Single Oral Dose of PF-07081532 20 mg in Participants With Varying Degrees of Renal Impairment
Description: Plasma Cmax was observed directly from data.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1
Population: Pharmacokinetic (PK) parameter set included all participants who received at least 1 dose of PF-07081532 and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 5 | 8
Nanograms per milliliter (ng/mL) | 2084 (50) | 1823 (24) | 1978 (30)

2. Primary Outcome: Unbound Cmax (Cmax,u) for PF-07081532 Following a Single Oral Dose of PF-07081532 20 mg in Participants With Varying Degrees of Renal Impairment
Description: Cmax,u was calculated as fu*Cmax. Plasma Cmax was observed directly from data. fu was defined as the fraction of unbound drug in plasma, and was obtained from measurement of protein binding.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1
Population: PK parameter set included all participants who received at least 1 dose of PF-07081532 and had at least 1 of PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 5 | 8
ng/mL | 0.6178 (44) | 0.5895 (17) | 0.8239 (27)

3. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) for PF-07081532 Following a Single Oral Dose of PF-07081532 20 mg in Participants With Varying Degrees of Renal Impairment
Description: AUCinf was calculated as AUClast + (Clast*/kel). AUClast was defined as area under the plasma concentration-time profile from time 0 to the time last measurable concentration, and was calculated using linear/log trapezoidal method. Clast* was defined as the predicted plasma concentration at the last quantifiable time point estimated from log-linear regression analysis. kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1
Population: PK parameter set included all participants, who received at least 1 dose of PF-07081532, had at least 1 of PK parameters of interest calculated. Number of Participants Analyzed represents the number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hours/milliliter (ng*h/mL)
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 4 | 5 | 7
Nanograms*hours/milliliter (ng*h/mL) | 59820 (41) | 45600 (21) | 43870 (33)

4. Primary Outcome: Unbound AUCinf (AUCinf,u) for PF-07081532 Following a Single Oral Dose of PF-07081532 20 mg in Participants With Varying Degrees of Renal Impairment
Description: AUCinf,u was calculated as fu*AUCinf. AUCinf was calculated as AUClast + (Clast*/kel). AUClast was defined as area under the plasma concentration-time profile from time 0 to the time last measurable concentration, and was calculated using linear/log trapezoidal method. Clast* was defined as the predicted plasma concentration at the last quantifiable time point estimated from log-linear regression analysis. kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. fu was the fraction of unbound drug in plasma, and was obtained from measurement of protein binding.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 4 | 5 | 7
ng*h/mL | 17.51 (56) | 14.75 (31) | 18.44 (35)

5. Primary Outcome: Unbound Fraction (fu) for PF-07081532 Following a Single Oral Dose of PF-07081532 20 mg in Participants With Varying Degrees of Renal Impairment
Description: fu was the ratio of unbound drug concentration to the total drug concentration, and was obtained from measurement of protein binding.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 15, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 5 | 8
Ratio | 0.0002964 (14) | 0.0003234 (15) | 0.0004163 (15)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Treatment-emergent AEs (TEAEs) = AEs occurred after starting of study treatment and up to the end of study that were absent before treatment or that worsened relative to pretreatment state. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-related AEs and SAEs were determined by the investigator. Severe=an event that prevents normal everyday activities.
Time Frame: From time of administration of study treatment on Day 1 up to the end of the study (up to a maximum of 31 days post dose)
Population: Safety analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 5 | 8
Participants
  Participants With All-Causality TEAEs | 1 | 2 | 1
  Participants With All-Causality SAEs | 0 | 0 | 0
  Participants With All-Causality Severe TEAEs | 0 | 0 | 0
  Participants With Treatment-Related TEAEs | 0 | 2 | 0
  Participants With Treatment-Related SAEs | 0 | 0 | 0
  Participants With Treatment-Related Severe TEAEs | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Parameters analyzed for lab examination included hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin [MCH], MCH concentration, platelet count, white blood cell count, absolute [Abs] total neutrophils, Abs eosinophils, Abs monocytes, Abs basophils, Abs lymphocytes), chemistry (Scr, Scys, fasting plasma glucose, calcium, sodium, potassium, chloride, magnesium, phosphate, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma glutamyl eGFR), urinalysis (pH, qualitative [qual] glucose, qual protein, qual blood, ketones, nitrites, leukocyte, esterase, urobilinogen, urine bili, microscopy). Lab parameters meeting the predefined criteria and with at least 1 occurrence from baseline up to end of study are reported. Baseline was defined as the last pre-dose measurement.
Time Frame: Pre-dose, 72 and 144 hours post dose on Day 1
Population: Safety analysis set included all participants assigned to study intervention who took at least 1 dose of study intervention. Number of Participants Analyzed represents the total number of participants who were evaluable for this outcome measure. Number Analyzed for each lab parameter represents the number of participants who had at least 1 post dose measurement for the parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 4 | 5 | 8
Participants
  Hematology-Hemoglobin (grams per deciliter [g/dL])<0.8*lower limit of normal (LLN) | 0 | 1 | 4
  Hematology-Hematocrit (%)<0.8*LLN | 0 | 0 | 4
  Hematology-Erythrocytes (10^12/Liter [L])<0.8*LLN | 0 | 1 | 4
  Hematology-Eosinophils (10^9/L)>1.2* upper limit of normal (ULN) | 0 | 0 | 1
  Clinical Chemistry-Gamma Glutamyl Transferase (units [U]/L)>3.0*ULN | 0 | 0 | 1
  Clinical Chemistry-Urea Nitrogen (milligrams [mg] / dL)>1.3*ULN | 1 | 4 | 7
  Clinical Chemistry-Creatinine (mg/dL)>1.3*ULN | 0 | 3 | 8
  Clinical Chemistry-Urate (mg/dL)>1.2*ULN | 0 | 0 | 1
  Clinical Chemistry-Potassium (milliequivalents [mEq] / L)>1.1*ULN | 0 | 0 | 1
  Clinical Chemistry-Magnesium (mg/dL)<0.9*LLN | 0 | 1 | 0
  Clinical Chemistry-Phosphate (mg/dL)<0.8*LLN | 0 | 0 | 1
  Clinical Chemistry-Phosphate (mg/dL)>1.2*ULN | 0 | 1 | 0
  Clinical Chemistry-Bicarbonate (mEq/L)<0.9*LLN | 0 | 0 | 1
  Clinical Chemistry-Fasting Glucose (mg/dL)>1.5*ULN | 1 | 3 | 2
  Urinalysis-Urine Glucose Positive: number analyzed (Participants) | 4 | 5 | 6
  Urinalysis-Urine Glucose Positive | 0 | 1 | 1
  Urinalysis-Urine Protein Positive: number analyzed (Participants) | 4 | 5 | 6
  Urinalysis-Urine Protein Positive | 0 | 2 | 5
  Urinalysis-Urine Hemoglobin Positive: number analyzed (Participants) | 4 | 5 | 6
  Urinalysis-Urine Hemoglobin Positive | 0 | 0 | 1
  Urinalysis-Nitrite Positive: number analyzed (Participants) | 4 | 5 | 6
  Urinalysis-Nitrite Positive | 1 | 0 | 1
  Urinalysis-Leukocyte Esterase Positive: number analyzed (Participants) | 4 | 5 | 6
  Urinalysis-Leukocyte Esterase Positive | 1 | 1 | 2

8. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-Defined Categorical Criteria
Description: Vital signs including single, seated blood pressure (BP) and pulse rate were measured with the participant's arm supported at the level of the heart, and recorded to the nearest mmHg, following a seated rest of ≥5 minutes. Same arm (preferably the dominant arm) was used for BP/pulse rate assessment throughout the study. Vital signs meeting the predefined criteria and with at least 1 occurrence from baseline up to end of study are reported. Baseline was defined as the last pre-dose measurement.
Time Frame: At admission on Day -1, pre-dose, and 24, 72, and 144 hours post the dose on Day 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 5 | 8
Participants
  Systolic BP (mm Hg) Increase >=30 mm Hg: number analyzed (Participants) | 5 | 5 | 6
  Systolic BP (mm Hg) Increase >=30 mm Hg | 0 | 1 | 1
  Diastolic BP (mm Hg) Increase >=20 mm Hg | 0 | 0 | 1
  Diastolic BP (mm Hg) Decrease >=20 mm Hg | 0 | 0 | 1

9. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-Defined Categorical Criteria
Description: Supine standard 12-lead ECGs utilizing limb leads (with a 10-second rhythm strip) were collected at times specified in the time frame using an ECG machine that automatically calculates the HR and measures PR interval, QT interval, QTcF, and QRS complex. All scheduled ECGs were performed after the participant had rested quietly for at least 5 minutes in a supine position. ECG data meeting the predefined criteria and with at least 1 occurrence from baseline up to end of study were reported. Baseline was defined as the last pre-dose measurement.
Time Frame: Pre-dose, and 144 hours post the dose on Day 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 5 | 5 | 8
Participants | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: From time of administration of study treatment on Day 1 up to the end of the study (up to a maximum of 31 days post dose).
Description: Total number at risk below refers to the number of participants evaluable for AEs. All adverse events are reported, whether or not considered related to the study intervention.
Arm/Group | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 1/5 | 2/5 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild Renal Impairment (N=5) | Moderate Renal Impairment (N=5) | Severe Renal Impairment (N=8)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to the termination of clinical development of PF-07081532, and no participants without renal impairment were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT05510245/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT05510245/SAP_001.pdf